CLINICAL TRIAL: NCT04940819
Title: A Mobile Application Based Dietary Self Management Intervention in Chinese Chronic Kidney Disease Patients: a Multi-Center Randomized Controlled Study
Brief Title: A Mobile Application Based Dietary Self Management Intervention in Chinese Chronic Kidney Disease Patients
Acronym: CRISS-MADE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Limeng Chen, Director, Department of Nephrology, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRISS-Diet
Record Dates: First submitted 2021-05-31; First posted 2021-06-28 (Actual); Last update posted 2021-06-28 (Actual); Status verified 2021-06

CONDITIONS: Chronic Renal Disease
Keywords: Chronic Renal Disease; Dietary Management; Mobile Application
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobile Application Intervention (Experimental): Participants in this arm will receive mobile application dietary intervention as well as usual CKD dietary care.
  Interventions: Behavioral: Mobile Application for Dietary Management
- Care as Usual (No Intervention): Participants in this arm will receive usual CKD dietary care.

INTERVENTIONS:
Behavioral: Mobile Application for Dietary Management — A mobile application developed by a multi-disciplinary team will be used in the dietary management of CKD patients. The application is patient orientated. It has 4 core features including food searching, dietary logging, personalized key nutrient intake feedback and patient-caregiver interaction.
  Arms: Mobile Application Intervention

SUMMARY:
This is a multi-center randomized controlled study. This study aims to investigate the acceptability and efficacy of a newly developed mobile application in the dietary management of chronic kidney disease (CKD) patients.

DETAILED DESCRIPTION:
The prevalence of CKD has reached 10.8% in China. Increasing in prevalence of other non-communicable disease such as hypertension, diabetes and obesity is contributing to this rise in CKD and end-stage renal disease prevalence. Diet is a strong modifiable factor in these diseases. Dietary control is also an integral part in CKD disease self management. However, the complexity in the dietary management of CKD makes it hard for patients to adequately self manage. With the development of smart phone, many mobile applications have been developed to suit the need of patients with chronic diseases. But there has been a scarce of randomized trial to support the feasibility, acceptability and efficacy of these mobile applications.

Our study aims to employ a newly developed dietary logging and monitoring application in the primary care setting of CKD patients to test its acceptability and efficacy in disease control.

The application is developed by a multidisciplinary team in a tertiary care center. The main features include searching and logging foods, receiving realtime feedback on key nutrient intake levels and facilitating patient-care giving communication.

We plan to enroll 14 tertiary hospitals and 42 secondary hospitals in 7 geographical regions in China aiming to reach participants in resource poor areas. Participants will be randomized with 1 to 1 ratio to either receiving mobile application dietary intervention or usual dietary consultation. The planned intervention period is 3 months. We will monitor biochemical parameters relating to dietary control and evaluate patient-centered outcomes concerning CKD self management and control.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with CKD for more than 3 months
* Objective measures of kidney disease (fulfill one of the following): 1) eGFR≤60ml/min/1.73m^2; 2) Proteinuria (Protein + on dipstick or 24 hour urine protein>0.3g or albumin-to-creatinine ratio (ACR) >30mg/mmol or protein-to-creatinine ratio (PCR) >50mg/mmol); 3) Imaging proven kidney disease (Atrophy, stone formation, cystic kidney disease, or other structural abnormality)
* Having access to a mobile phone and is capable of using the dietary intervention application

Exclusion Criteria:

* Can not provide history of kidney disease or can not provide laboratory result for the past 3 month
* Can not use a mobile phone or deemed unfit to participate by their treating nephrologist

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9863 (Estimated)
Dates: Start 2021-06 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Dietary Intake | 3 months
  Dietary intake of calorie, protein, sodium, potassium and phosphate evaluated by three-day diet records (3DDR)
Diet Quality | 3 months
  Calculated by Chinese Healthy Eating Index
Blood Pressure | 3 months
  Measure BP in office visits after the intervention period. Changes in antihypertensive medication requirements (total number, dose, class) will be collected from participants and verified with hospital records.
change in estimated Glomerular Filtration Rate (eGFR) | 3 months
  blood draw (fasting) before and after intervention period
Change in Proteinuria | 3 months
  spot urine before and after intervention period
Change in Disease Related Quality of life | 3 months
  Measured by Kidney Disease Quality of Life 36-Short Form questionnaire
Change in Self-Efficacy for Managing Chronic Disease Scale | 3 months
  Score of Self-Efficacy for Managing Chronic Disease Scale (6 items, each measured on a 1-10 likert scale, higher score indicate better self-efficacy) before and after intervention period
Change in Perceived Medical Condition Self-Management Scale (PMCSMS） | 3 months
  Measured by Perceived Medical Condition Self-Management Scale (8-item CKD-specific version of the PMCSMS, each item is scored on a 1-5 likert scale, with higher score indicating better self management on item 3/4/5/8 and lower score indicating better self management on item 1/2/6/7) before and after intervention

SECONDARY OUTCOMES:
Blood Chemistry (Potassium, Bicarbonate, Phosphate) | 3 months
  blood draw (fasting) before and after intervention period
Urine Sodium/potassium Ratio | 3 months
  Measured by spot urine at baseline and after intervention
Salt Taste Threshold | 3 months
  Salt taste threshold measured using salt-impregnated test strips before and after the intervention period
Kidney Nutrition Knowledge, Attitude and Practice | 3 months
  Measured by self developed questionnaire about knowledge, attitude and practice in kidney disease specified diet
Acceptability of the Application | 3 months
  Measured by user acceptability survey and semistructured interviews conducted in participants and nephrologists
Adherence | 3 months
  Total number of diet diary logged by participants over complete study period (more than 60% logged is deemed good adherence)
Adoption | 3 months
  Measured by percentage of complete dietary log in days will be counted (>1200kcal deemed as complete log)
Change in the score of Generalized Anxiety Disorder Scale | 3 months
  Measured by Generalized Anxiety Disorder Scale (a 7-item self-report scale. Items are rated on a 4-point Likert-scale with 0 = not at all to 3 = nearly every day ) before and after intervention
Change in the score of Hospital Anxiety and Depression Scale | 3 months
  Measured by Hospital Anxiety and Depression Scale (14 items each rated on a 0-3 score, with higher score indicating worse anxiety or depression symptoms) before and after intervention

OTHER OUTCOMES:
Change in Chronic Kidney Disease Self-Efficacy Instrument | 3 months
  Score of Chronic Kidney Disease Self-Efficacy Instrument before and after intervention period
Change in Kidney Disease Behaviors Inventory | 3 months
  Kidney Disease Behaviors Inventory before and after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Limeng Chen, MD, PhD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang L, Wang F, Wang L, Wang W, Liu B, Liu J, Chen M, He Q, Liao Y, Yu X, Chen N, Zhang JE, Hu Z, Liu F, Hong D, Ma L, Liu H, Zhou X, Chen J, Pan L, Chen W, Wang W, Li X, Wang H. Prevalence of chronic kidney disease in China: a cross-sectional survey. Lancet. 2012 Mar 3;379(9818):815-22. doi: 10.1016/S0140-6736(12)60033-6. PMID 22386035
- [Background] Stevenson JK, Campbell ZC, Webster AC, Chow CK, Tong A, Craig JC, Campbell KL, Lee VW. eHealth interventions for people with chronic kidney disease. Cochrane Database Syst Rev. 2019 Aug 6;8(8):CD012379. doi: 10.1002/14651858.CD012379.pub2. PMID 31425608
- [Background] Lim JH, Lim CK, Ibrahim I, Syahrul J, Mohamed Zabil MH, Zakaria NF, Daud ZAM. Limitations of Existing Dialysis Diet Apps in Promoting User Engagement and Patient Self-Management: Quantitative Content Analysis Study. JMIR Mhealth Uhealth. 2020 Jun 1;8(6):e13808. doi: 10.2196/13808. PMID 32478665